CLINICAL TRIAL: NCT06940362
Title: Changing Youth Narratives on Firearm Violence: A Community Collaborative Intervention - Phases 1 and 2
Brief Title: Changing Youth Narratives on Firearm Violence ("Run It Up") Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCR234833
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Injury Prevention
Keywords: Community intervention, quasi-experimental design, youth firearm violence prevention

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design, with intervention and comparison community
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth intervention arm (Experimental): Training and mentoring of 12-16 year old youth in non-violent personal/career trajectories, supported by a social media campaign and a community steering committee.
  Interventions: Behavioral: Changing narrative intervention modules

INTERVENTIONS:
Behavioral: Changing narrative intervention modules — Training and mentoring of 12-16 year old youth in non-violent personal/career trajectories, supported by a social media campaign and a community steering committee.

SUMMARY:
The Run It Up project is an experimental, theory-driven effort to address a specific connection between structural factors, youth identity development, and violence, where structural factors in some communities may limit adolescent beliefs about potential life-trajectories ("possible selves"), and foreground potential trajectories that include violence as integral. The intervention seeks to counter that dynamic by: 1) identifying alternative, non-violent identity trajectories that have attributes meaningful for youth and actualizing those trajectories through a community support structure; and 2) developing and disseminating multiple media products featuring narratives about these alternative trajectories. The goal is to change the calculation of possible selves for adolescents in the identity development stage through the introduction, and actualization, of desirable, tangible trajectories that do not involve violence or pro-violence norms, resulting in a reduction of youth involvement in firearm violence. The intervention and research is being conducted through a partnership between the George Washington University Milken Institute School of Public Health and the Washington, DC community of Washington Highlands, and is funded through a grant from the National Institute on Minority Health and Health Disparities (NIMHD). In the first phase, formative research was completed to identify attributes and alternative non-violent trajectories, determine intervention elements, develop an intervention "brand" representing the attributes, develop a baseline-follow-up survey measuring theoretical mediators/moderators, outcomes, and other potential influencing factors, and identify community data to be used for a time-series analysis. Now in the second phase, the baseline data from a sample of community youth and parents/guardians are currently being collected prior to implementing the intervention. Evaluation is a two group, quasi-experimental community cohort design using survey and community-level data.

DETAILED DESCRIPTION:
The overall design for the intervention evaluation is a two group, quasi-experimental community cohort design with a pretest (baseline) and multiple post-tests (follow-ups). A baseline survey and two follow-ups of 12-16-year-old youth and one parent/guardian per youth will be collected in the intervention and comparison communities, separately measuring a number of resilience, risk-related and demographic variables, hypothesized mediators/moderators linked to the intervention and its theory of change, intervention and related media exposure, and self-report outcomes. The comparison community (Marshall Heights) has been matched to the intervention community (Washington Highlands) as closely as possible on demographic and violence data (e.g., 95% African American in the intervention community, vs 90% African American in the comparison community; both communities have high poverty rates). A preliminary analysis will be conducted at each follow-up, with full analysis after the last follow-up. The research team will also collect firearm and related violence data as well as place-based aggregated data from designated community Census tracts for two years pre-intervention to the final intervention year for both communities, either monthly or quarterly, depending on whether there are enough samples in each period, in order to conduct interrupted time series analysis (ITSA) to assess the intervention effect on community-level outcomes.

Sampling Because there is no sampling frame from which to randomize, the research team is using a targeted snowball method through community partners (the CSC) who are familiar with most community families. Recruitment will occur through these interpersonal networks, using flyers with study information and eligibility requirements, prompting a snowball process where initial contacts recruit others. This method is more productive, facilitates the consent-assent process and recruitment of parents/guardians, and may avoid inherent safety concerns compared to sending staff to knock on doors for recruitment. Further, it will likely increase awareness and trust in the effort. It will also support a community cohort design, in which the same samples are followed up over time, with an improved ability to make causal inferences.

To increase rigor, the annual survey sample size proposed in the funding application has been increased from 200 youth/200 parents to 250 youth and the same number of parents (in both communities, for a total n of 500 youth, 500 parents each wave), in order to achieve enough power in the supplemental propensity score analyses, and for dose-response analyses. Along with that, the research team (including the community partners) will implement recruiting strategies to maximize direct youth participation in the intervention activities, to reach a goal of approximately 100-150 youth participating in the intervention activity tracks. These participants assessed at baseline will be followed up at 12 and 24 months after the baseline survey, separately.

Administration The baseline and follow-up surveys will be administered via mobile phone and tablets to a community sample of youth and parents/guardians. In the intervention community, data collection will not be limited to youth who participate in the alternative trajectory intervention activity tracks, because the goal is to assess intervention effects on community youth as a whole (including those directly participating in activities). However, to improve linkage between survey data and actual intervention participants, survey and intervention participant IDs will be linked by participant names, which will be maintained in a separate password-protected secure file and not appear on any survey or intervention process data. Variables will be created indicating dose to intervention exposure including participation in the intervention activity tracks and " and "media exposure". In this way, it will be possible to assess the dose-response effect among the youth in the intervention community. The survey and data storage will use REDCap software for security and efficiency.

Process and Qualitative Measures Extensive process data will be collected, e.g. attendance of each session and satisfaction with the session for each youth participating in the intervention activity tracks. In addition, each program year, 15 youth who are involved in any program activities will be randomly selected for a one-hour interview about experiences with program media/messaging and any perceived changes resulting from this exposure. The research team will also conduct interviews with two adults named by the youth as program-related influencers or mentors, to assess any changes mentors have seen in the youth, and perceptions of factors leading to the changes. These qualitative interviews (n=45) in Years 3-5 will be conducted and analyzed using the same methods outlined for the Phase One formative research.

Analyses Originally planned analyses include descriptive analyses, Difference-in-Difference (DID) analysis to test intervention effect, sensitivity analysis to assess contamination, mediation analysis and moderation analyses based on survey data, and interrupted time series analysis (ITSA) based on community data. A number of changes have been made in the original analytical plan to increase rigor, recognizing the complexity of a quasi-experimental design with one intervention and one comparison community. First, the interrupted time series component has been strengthened in several ways. This component entails tracking a set of data at the community level that we would expect to change (in a positive direction) over time as a result of the intervention. As a minimum set of community data, each occurrence of any crime, gun-related crime, non-gun-related crime in the study Census tracts will be derived from data reported through the website crimecards.dc.gov, tracked monthly from two years before the intervention and then across the intervention period. The data will be aggregated over time and over the specific Census tracts in each community (by matching addresses to Census tract) to calculate monthly or quarterly crime rate (number of crimes divided by the population), depending on how many crimes in each community per month. In addition, the research team is seeking community-level placebo measures that will not be changed by the intervention. These will most likely include: (1) Temporary Assistance for Needy Families (TANF) data from the DC Department of Health; and (2) child poverty data from the DC Office of Planning -- across time in each Census tract and then aggregated for analysis. The ITSA with placebo outcomes will increase the robustness in the analyses. Similarly, for DID using survey data, placebo measures have been added to the survey that are not expected to change as a result of the intervention - for example, diet, or self-reported height and weight -- as an additional means to test the robustness of DID.

In addition, propensity score matching has been added as a supplemental analysis. For this, youth will be matched based on their baseline characteristics (sociodemographic and outcome variable at baseline) from the intervention community and comparison community to mimic an RCT for assessment of the intervention effect. Propensity score analysis will be implemented with "teffect psmatch" using STATA software.

Finally, the research team is collecting survey IDs, participant IDs, and tracking short-term outcome and process data collected by intervention component, social media/community event exposure, and brand equity data , allowing for analysis of intervention effect by type and degree of exposure - because it will be possible to link participant IDs and survey IDs.

ELIGIBILITY:
Inclusion Criteria:

• Resident of intervention community, within age limits

Exclusion Criteria:

• Not resident of intervention community, outside of age limits

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-11-07 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in youth firearm violence involvement | 2 1/2 years
  Change in self-reported violence involvement by participants (via survey) and changes in community violence data (incidence, from police and health tracking data).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Edberg, PhD, MA, Principal Investigator — George Washington University
Locations (1):
- George Washington University Milken Institute School of Public Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Results will only be reported in the aggregate, with no individual identifiers.

REFERENCES:
- [Background] Sokol R, Walton M, Lee D, Seewald L, Del Toro VM, Farooqui M, Sallabank G, Zimmerman M, Edberg M, Wang Y, Zakrison T, Tung EL, Hillegass WB, Vearrier L, Zhang L, Kutcher ME, Blachman-Demner D, Carter PM. Advancing Science to Prevent Firearm Violence in Communities: A Process for Harmonizing Studies to Develop Research Infrastructure. Prev Sci. 2024 Oct;25(7):1122-1132. doi: 10.1007/s11121-024-01723-5. Epub 2024 Sep 20. PMID 39304578
- [Background] Edberg MC, Cleary SD, Andrade EL, Evans WD, Quinteros-Grady L, Alvayero RD, Gonzalez A. The Adelante project: Realities, challenges and successes in addressing health disparities among central American immigrant youth. Cultur Divers Ethnic Minor Psychol. 2022 Jul;28(3):402-412. doi: 10.1037/cdp0000368. Epub 2021 Dec 23. PMID 34941282
- [Background] Edberg M. The cultural persona as nexus between structural marginalization and youth risk behavior. J Community Psychol. 2020 Sep;48(7):2138-2155. doi: 10.1002/jcop.22368. PMID 32841383